CLINICAL TRIAL: NCT06232720
Title: Q300 User Site Testing Study
Brief Title: User Site Testing Study to Evaluate Usability of the Q300™ Device Under "Real-life Conditions" in a Reproductive Laboratory Environment Use
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: QART Medical (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Q300-02
Record Dates: First submitted 2023-07-03; First posted 2024-01-31 (Actual); Last update posted 2024-01-31 (Actual); Status verified 2024-01

CONDITIONS: to Aid in Sperm Selection for ICSI

STUDY DESIGN:
Intervention Model Description: The study will be an open label study, non-controlled and non-randomized.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Q300 QART Medical — The Q300TM Imaging system includes a Quantitative Phase Microscope. Q300TM uses a low intensity coherent light source, in a uniquely configured interferometer, which measures light delay as it passes different locations across the sperm cell. The amount

SUMMARY:
User Site Testing Study to evaluate usability of the Q300™ device under "real-life conditions" in a reproductive laboratory environment use.

DETAILED DESCRIPTION:
Testing the Usability of the Q300™ device.

Specific objectives of this evaluation are as follows:

* Confirm the comprehensiveness of the User Manual in providing adequate instructions for proper system operation and application.
* Assist in further improving the User Manual and generate input to Manufacturer on way to improve the Q300™ device.
* Demonstrate that Q300 can be used by the intended users without use errors or problems that negatively impact system use.
* Evaluate the effect of using the Q300™ on the user's (i.e. embryologist's) ability to prospectively select morphologically-compliant sperm cells.
* Assist in determining the inclusion/exclusion criteria for subsequent clinical investigations.
* Further improve the QART Feature Extraction algorithm observing general morphological phenotypes in sperm cells.
* Evaluate effect of using the Q300 on the clinical outcome

ELIGIBILITY:
Inclusion Criteria:

* Patient intended for ICSI recruited from the hospital's IVF (both male and female are considered patients in this study).
* Male, Age >18 yrs
* Female age < 40 yrs
* Patients signed informed consent prior study procedures.
* Fresh Oocytes
* Fresh ejaculated motile sperm and presence of motile sperm at the time of sperm selection for ICSI
* Fresh oocytes
* Non severe male factor (TMC>1*10^6/mL)
* Unexplained factor infertility
* AFC >=13mm during ovarian stimulation prior to ovulation trigger or induction#>=5 in the cycle

Exclusion Criteria:

* Frozen spermatozoa
* Immotile sperm
* Severe Oligozoospermia (less than 1 million sperm cells after preparation).
* Spermatozoa extracted by TESA/ TESE
* Frozen oocytes
* Egg or ovulatory female factor such as low ovarian reserve (menstrual cycle, per AFC. AMH test- if performed) or non-typical eggs or eggs with severe pathology (qualitative; please find
* That the instructions for use of Q300TM have not been fully followed (poor quality of images etc…)
* Inability to reliably trace sperm-oocyte-embryo clinical outcome throughout the process.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Estimated)
Dates: Start 2024-02-15 (Estimated); Primary Completion 2025-01-31 (Estimated); Study Completion 2025-03-15 (Estimated)

PRIMARY OUTCOMES:
Usability | 1 year
  Usability surveys to users including user manual comprehensiveness questionnaire (evaluation of critical steps in the procedure, correct use, feedback on training provided).
Usable blastocyst formation rate | 5 days
  Number of usable (transferred or frozen) embryos per cycle (Gardner 2BB at day 5 or equivalent or grade "good" according to Istanbul consensus for cleavage-stage.

CONTACTS AND LOCATIONS:
Overall Officials: Orly Schwartz, Study Director — QART Medical
Locations (1):
- Barzilay Medical Center, Ashkelon, Israel

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Michailov Y, Amsalem E, Umanski N, Tamadaev V, Friedler S, Saar-Ryss B. Clinical outcome using the Q300 device in a reproductive laboratory environment: an open-label, non-controlled and non-randomized study. Reprod Biol Endocrinol. 2025 Jun 10;23(1):90. doi: 10.1186/s12958-025-01424-w. PMID 40495170
- [Derived] Michailov Y, Friedler S, Saar-Ryss B. First clinical pregnancy and delivery achieved after using a new 3D imaging technology for sperm selection: a case report. Front Reprod Health. 2025 Mar 7;7:1559684. doi: 10.3389/frph.2025.1559684. eCollection 2025. PMID 40124653